CLINICAL TRIAL: NCT00705705
Title: Targeted Social Network HIV Prevention Intervention
Brief Title: Effectiveness of an HIV Prevention Program That Targets the Inner Workings of High-risk Social Networks
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Yuri A. Amirkhanian, PhD, Associate Professor of Psychiatry and Behavioral Medicine, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: R01MH070316 (NIH); R01MH070316 (NIH); DAHBR 9A-ASPQ
Record Dates: First submitted 2008-06-24; First posted 2008-06-26 (Estimated); Last update posted 2011-11-11 (Estimated); Status verified 2011-11

CONDITIONS: HIV Infections
Keywords: High-Risk Behavior; Men Who Have Sex With Men; HIV Seronegativity
MeSH Terms: conditions — HIV Infections; Homosexuality

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Participating social networks will receive standard HIV risk-reduction counseling and network leadership training on HIV prevention.
  Interventions: Behavioral: Network leader training; Behavioral: Standard HIV risk-reduction counseling
- 2 (Active Comparator): Participating social networks will receive standard HIV risk-reduction counseling.
  Interventions: Behavioral: Standard HIV risk-reduction counseling

INTERVENTIONS:
Behavioral: Network leader training — Network leaders will receive a nine-session training segment designed to enable them to motivate their peer networks to reduce sexual risk. The sessions will teach the identified leader of each network how to communicate HIV prevention messages to other members of his or her personal social network. Leaders will be asked to share these messages with other members of their groups.
  Arms: 1
Behavioral: Standard HIV risk-reduction counseling — Participants will undergo interviews about their friendship groups, sexual behavior, substance abuse, STD treatment history, condom use, and beliefs about HIV/AIDS. Participants will undergo a brief session about HIV/AIDS prevention methods after the first interview.

SUMMARY:
This study will determine whether an HIV prevention program that targets the inner workings of social networks at high risk for HIV and other sexually transmitted diseases is effective in reducing frequency of high-risk sexual behaviors among network members.

DETAILED DESCRIPTION:
Over the past decade, the number of new HIV infections in the United States has remained on a steady level, with approximately 40,000 Americans contracting the disease each year. Risk of contracting HIV is not evenly distributed throughout the population, with groups such as intravenous drug users, men who have sex with men (MSM), and impoverished people in inner cities being disproportionately affected. Many members of these groups have already made risk-reduction behavior changes, but there are certain clusters or networks of people within these populations who remain at a greater risk of HIV infection and who account for the majority of new infections. Therefore, more effective HIV prevention approaches directed toward high-risk social networks are needed. Training social leaders within the high-risk networks to communicate HIV prevention messages directly to their members may be an effective means of reaching these vulnerable population segments. This study will evaluate the effectiveness of an HIV prevention program that targets the inner workings of high-risk social networks (particularly young MSM and young high-risk heterosexual adult men and women) in reducing frequency of risky sexual behaviors among network members.

Participation in this study will last up to 2 years and will include the leaders and general members of multiple social networks. First, the eligibility of a given social network will be determined through a period of in-depth formative ethnographic research that will include a 20-minute interview with members of the social networks. During the eligibility interview, participants will be asked to provide personal information about themselves and their close friends, called a friendship group in this study. After the interview, participants will be asked to distribute a flyer about participating in the study to their friendship group. If enough members of the friendship group agree to complete the initial interview and the group meets the eligibility criteria, then members of the group will be asked to participate in the assessment interviews.

The first 1-hour assessment interview will be conducted at baseline and will include two parts. During the first part of the interview, participants will complete a survey about the friendship group, including questions about their most and least trusted members and communication among group members. The second part of the interview will include taking a computer survey with questions about sexual behavior, substance abuse, STD treatment history, condom use, and beliefs about HIV/AIDS. After completing the interview, participants will undergo a brief HIV/AIDS prevention counseling session. Participants will repeat this assessment interview 12 and 24 months later.

When at least half of the friendship group has completed the first assessment interview, the group will be assigned randomly to one of two conditions:

* For groups assigned to Condition 1, participants will receive a phone call when it is time for their repeat assessment interviews. In addition, a computer program will identify one person as the leader of the friendship group, and this person will be asked to attend nine 3-hour meetings over 17 weeks. These meetings will train and encourage leaders to provide positive HIV/AIDS prevention advice to the members of their friendship group.
* For groups assigned to Condition 2, participants will receive a phone call when it is time for their repeat assessment interviews. If the leadership program in Condition 1 appears to be effective, participants may be offered the same program at a later time.

Study participation will be complete after the 24-month assessment interview.

ELIGIBILITY:
Inclusion Criteria:

* Identified by the network leader as a member of the social group (e.g., men who have sex with men, young heterosexual men and women)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 852 (Actual)
Dates: Start 2004-07; Primary Completion 2009-03 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Frequency of high-risk sexual practices | Measured at baseline and Months 12 and 24

SECONDARY OUTCOMES:
Effectiveness and usefulness of HIV prevention intervention as a public health approach for reaching population segments that remain vulnerable to HIV and other STDs | Measured at baseline and Months 12 and 24

CONTACTS AND LOCATIONS:
Overall Officials: Yuri A. Amirkhanian, PhD, Principal Investigator — Medical College of Wisconsin; David W. Seal, PhD, Study Director — Medical College of Wisconsin; Jeffrey A. Kelly, PhD, Study Director — Medical College of Wisconsin; Carol L. Galletly, JD, PhD, Study Director — Medical College of Wisconsin; Laura R. Glasman, PhD, Study Director — Medical College of Wisconsin; Timothy L. McAuliffe, PhD, Study Director — Medical College of Wisconsin
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States